CLINICAL TRIAL: NCT01552772
Title: An Open-label, Safety and Tolerability Trial of Aripiprazole IM Depot Treatment Initiation in Adult Subjects With Schizophrenia Stabilized on Atypical Oral Antipsychotics Other Than Aripiprazole
Brief Title: Safety and Tolerability Trial of Aripiprazole IM Depot Treatment in Adult Subjects With Schizophrenia Stabilized on Oral Antipsychotics Other Than Aripiprazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-11-289
Record Dates: First submitted 2012-02-13; First posted 2012-03-13 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Schizophrenia
Keywords: Safety; Tolerability; Schizophrenia; Aripiprazole
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole IM Depot (Experimental)
  Interventions: Drug: Aripiprazole IM Depot

INTERVENTIONS:
Drug: Aripiprazole IM Depot — 400 mg intramuscular injection of aripiprazole
  Other Names: Abilify

SUMMARY:
This study will test the safety of an aripiprazole injection in subjects with schizophrenia that are currently taking oral antipsychotic medication other than aripiprazole. Subjects in this study will receive one injection of aripiprazole and will need to stop taking their other antipsychotic medication two weeks after the injection. The study will last one month. Subjects will be required to come to a clinic for evaluations and drug and urine collection five times during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female individuals between 18 and 64 years of age, inclusive, with a diagnosis of schizophrenia as defined by DSM-IV-TR criteria.
2. Good physical health as determined by no clinically significant deviation from normal in medical history, clinical laboratory determination, ECGs, or physical examinations.
3. Ability to provide written informed consent or consent obtained from a legally acceptable representative (as required by IRB) prior to the initiation of any protocol-required procedures.
4. Body mass index of 18 to 35 kg/m2, inclusive.
5. Prior history of tolerating aripiprazole.
6. Subjects must be treated with one of the following atypical oral antipsychotic medications: risperidone, olanzapine, quetiapine, ziprasidone, or paliperidone and be clinically stable, per the investigator's judgment, for 14 days prior to the administration of aripiprazole IM depot

Exclusion Criteria:

1. Sexually active males who will not commit to utilizing 2 of the approved birth control methods or who will not remain abstinent during the trial and for 180 days following the last dose of trial medication, or have not had an orchidectomy or sexually active females of childbearing potential who will not commit to utilizing 2 of the approved birth control methods or who will not remain abstinent during the trial and for 150 days following the last dose of trial medication. Abstinence will be permitted if it is confirmed and documented at every trial visit. If employing birth control, 2 of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device, birth control pill, birth control depot injections, implant, condom or sponge with spermicide. Note: Women of childbearing potential (WOCBP) are defined as all women unless they have had an oophorectomy or hysterectomy or have been postmenopausal for 12 consecutive months.
2. Subjects who have met DSM-IV-TR criteria for substance abuse or dependence within the past 180 days; including alcohol and benzodiazepines, but excluding caffeine and nicotine. Subjects with a positive drug screen for cocaine or other drugs of abuse (excluding stimulants and other prescribed medications and marijuana).a
3. Subjects likely to require prohibited concomitant therapy during the trial, and use of any CYP2D6 and CYP3A4 inhibitors, or CYP3A4 inducers within 14 days prior to dosing and for the duration of the trial.
4. Females who are pregnant or lactating.
5. Subjects who had participated in any clinical trial involving a psychotropic medication within 1 month prior to enrollment; subjects who had participated in a previous IM depot trial within the last 6 months; or who had previously enrolled and received trial medication in an aripiprazole IM depot clinical trial.
6. Any major surgery within 30 days prior to enrollment.
7. Evidence of organ dysfunction or any clinically significant deviation from normal in physical, electrocardiographic, or clinical laboratory examinations.
8. Subjects who have a significant risk of committing suicide based on history or routine psychiatric status examination
9. Subjects currently in an acute relapse of schizophrenia.
10. Subjects with a current DSM-IV-TR diagnosis other than schizophrenia, including schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, amnestic or other cognitive disorders. Also, subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
11. Subjects who were considered treatment-resistant to antipsychotic medication. (Subjects needed to have shown a previous response to an antipsychotic medication other than clozapine.)
12. Subjects with a history of neuroleptic malignant syndrome or clinically significant tardive dyskinesia.
13. Subjects who are known to be allergic, intolerant, or unresponsive to prior treatment with aripiprazole or other quinolinones.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Wu, MD, Study Director — Otsuka Pharmaceutical Development and Commercialization
Locations (12):
- United States (12):
  - South Coast Clinical Trials, Anaheim, California
  - Comprehensive Clinical Development, Cerritos, California
  - Collaborative Neuroscience Network, Garden Grove, California
  - South Coast Clinical Trials, Norwalk, California
  - CNRI-San Diego, San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Comprehensive Clinical Development, Washington D.C., District of Columbia
  - Accurate Clinical Trials, Kissimmee, Florida
  - Compass Research, LLC, Orlando, Florida
  - St. Louis Clinical Trials, St Louis, Missouri
  - Community Clinical Research, Austin, Texas
  - Pillar Clinical Research, Dallas, Texas

REFERENCES:
- [Derived] Potkin SG, Raoufinia A, Mallikaarjun S, Bricmont P, Peters-Strickland T, Kasper W, Baker RA, Eramo A, Sanchez R, McQuade R. Safety and tolerability of once monthly aripiprazole treatment initiation in adults with schizophrenia stabilized on selected atypical oral antipsychotics other than aripiprazole. Curr Med Res Opin. 2013 Oct;29(10):1241-51. doi: 10.1185/03007995.2013.821973. Epub 2013 Jul 25. PMID 23822566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial to assess the safety and tolerability of aripiprazole intramuscular (IM) depot as an adjunctive therapy in adults with schizophrenia who were stabilized on any one of the atypical oral antipsychotics other than aripiprazole. In the United States, the trial was conducted in 60 enrolled participants and were screened in 12 centres.
Pre-assignment Details: The study consisted of a 30-day Screening period, a treatment phase of 28 days, and a Follow-up at 30 days after the last trial visit. Participants must have been stabilized on one of the following atypical oral antipsychotic medications for at least 14 days before Day 1: risperidone, quetiapine, olanzapine, ziprasidone, or paliperidone.
Groups:
- Aripiprazole IM Depot 400mg: Participants were stabilized on one of the following atypical oral antipsychotic medication for at least 14 days before Day 1: risperidone, quetiapine, olanzapine, ziprasidone, or paliperidone. On Day 1, participants were administered a single aripiprazole IM depot 400 mg injection. Concomitant to the aripiprazole IM depot injection, participants continued to receive their current atypical antipsychotic medication for 14 days.
Period: Overall Study
Arm/Group | Aripiprazole IM Depot 400mg
Started | 60
Completed | 56 (Participants who completed the Day 28 visit were defined as completers for the trial.)
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 1
Not completed — Protocol Deviation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aripiprazole IM Depot 400mg
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 (33.0)
  Male | 50 (67.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE).
Description: An AE was defined as any new medical problem, or exacerbation of an existing problem, experienced by a participant while enrolled in the trial, whether or not it was considered drug related by the study physician. A serious adverse event (SAE) was any untoward medical occurrence that resulted in death or was life-threatening or required inpatient hospitalization or prolonged hospitalization. TEAE stands for treatment emergent adverse events.
Time Frame: From the time the informed consent (ICF) was signed until follow-up at 30 days after the last trial visit (Day 28).
Population: The safety analyses dataset consisted of data from all enrolled participants who received one dose of trial medication, regardless of any protocol deviation. All observed data for these participants were included.
Measure: Number; unit: Participants
Arm/Group | Aripiprazole IM Depot 400mg
Number analyzed (Participants) | 60
Participants
  Participants with TEAE | 35
  Participants with serious TEAE | 1

2. Secondary Outcome: Change From Baseline in Total Score of Positive and Negative Syndrome Scale (PANSS) for Observed Cases (OC) Data.
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline, Week 1, 2, 4 and Last visit (Day 28).
Population: The efficacy analyses dataset consisted of enrolled participants who had at least one efficacy measurement. The OC dataset are participants who were evaluated at that visit on the efficacy variable under analysis (i.e. participants who had missing data due to drop out or other reasons were not included in the OC dataset).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400mg
Number analyzed (Participants) | 60
Units on a scale
  Week 1 (N= 59) | -2.42 (5.57)
  Week 2 (N= 56) | -2.86 (7.98)
  Week 4 (N= 57) | -3.82 (8.34)
  Last visit (N= 59) | -3.68 (8.26)

3. Secondary Outcome: Change From Baseline in Total Score of PANSS for Last Observation Carried Forward (LOCF) Data.
Description: as for outcome 2
Time Frame: Baseline, Week 1, 2 and 4
Population: The efficacy analyses dataset consisted of enrolled participants who have at least one efficacy measurement. The LOCF method was used to impute missing data at visits after Baseline for the efficacy analysis and for the safety extrapyramidal symptoms (EPS) assessment scales.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400mg
Number analyzed (Participants) | 60
Units on a scale
  Week 1 (N= 59) | -2.42 (5.91)
  Week 2 (N= 59) | -2.80 (7.83)
  Week 4 (N= 59) | -3.68 (8.26)

4. Secondary Outcome: Change From Baseline in PANSS Positive Sub-scale Score for OC Data.
Description: The Positive and Negative Syndrome Scale (PANSS) consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS positive subscale score was the sum of the rating scores for the 7 positive scale items from the PANSS panel. The 7 positive symptom constructs are delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline, Week 1, 2, 4 and Last visit (Day 28).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400mg
Number analyzed (Participants) | 60
Units on a scale
  Week 1 (N= 59) | -0.81 (2.45)
  Week 2 (N= 56) | -0.79 (3.37)
  Week 4 (N= 57) | -1.28 (2.89)
  Last visit (N= 59) | -1.25 (2.84)

5. Secondary Outcome: Change From Baseline in PANSS Positive Sub-scale Score for LOCF Data.
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS positive subscale score was the sum of the rating scores for the 7 positive scale items from the PANSS panel. The 7 positive symptom constructs are delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline, Week 1, 2 and 4
Population: The efficacy analyses dataset consisted of enrolled participants who have at least one efficacy measurement. The LOCF method was used to impute missing data at visits after Baseline for the efficacy analysis and for the safety EPS assessment scales.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400mg
Number analyzed (Participants) | 60
Units on a scale
  Week 1 (N= 59) | -0.81 (2.45)
  Week 2 (N= 59) | -0.78 (3.29)
  Week 4 (N= 59) | -1.25 (2.84)

6. Secondary Outcome: Change From Baseline in PANSS Negative Sub-scale Score for OC Data.
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS negative subscale score was the sum of the rating scores for the 7 negative scale items from the PANSS panel. The 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive apathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline, Week 1, 2, 4 and Last visit (Day 28).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400mg
Number analyzed (Participants) | 60
Units on a scale
  Week 1 (N= 59) | -0.78 (2.30)
  Week 2 (N= 56) | -1.14 (2.88)
  Week 4 (N= 57) | -0.96 (2.88)
  Last visit (N= 59) | -0.92 (2.84)

7. Secondary Outcome: Change From Baseline in PANSS Negative Sub-scale Score for LOCF Data.
Description: as for outcome 6
Time Frame: Baseline, Week 1, 2 and 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400mg
Number analyzed (Participants) | 60
Units on a scale
  Week 1 (N= 59) | -0.78 (2.30)
  Week 2 (N= 59) | -1.08 (2.82)
  Week 4 (N= 59) | -0.92 (2.84)

8. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity (CGI-S) Score in OC Data.
Description: The severity of illness for each participant was rated using the CGI-S scale. To assess CGI-S, the study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline, Week 1, 2, 4 and Last visit (Day 28).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400mg
Number analyzed (Participants) | 60
Units on a scale
  Week 1 (N= 59) | 0.02 (0.39)
  Week 2 (N= 56) | -0.09 (0.35)
  Week 4 (N= 57) | -1.14 (0.64)
  Last visit (N= 59) | -1.14 (0.63)

9. Secondary Outcome: Change From Baseline in CGI-S Score in LOCF Data.
Description: The severity of illness for each participant was rated using the CGI-S scale. To assess CGI-S, the rater or investigator answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline, Week 1, 2 and 4.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400mg
Number analyzed (Participants) | 60
Units on a scale
  Week 1 (N= 59) | 0.02 (0.39)
  Week 2 (N= 59) | -0.08 (0.34)
  Week 4 (N= 59) | -0.14 (0.63)

10. Secondary Outcome: Clinical Global Impression Improvement (CGI-I) Scale Score in OC Data.
Description: The efficacy of trial medication were rated for each participant using the CGI-I scale. The study physician must rate the participant's total improvement whether or not it is due entirely to drug treatment. All responses were compared to the participant's condition a baseline. Response choices include: 0 = not assessed; 1 =very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 =minimally worse; 6 = much worse; and 7 = very much worse.
Time Frame: Week 1, 2, 4 and Last visit (Day 28).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot 400mg
Number analyzed (Participants) | 60
Units on a scale
  Week 1 (N= 59) | 3.85 (0.45)
  Week 2 (N= 56) | 3.70 (0.57)
  Week 4 (N= 57) | 3.56 (0.78)
  Last visit (N= 59) | 3.58 (0.77)

11. Secondary Outcome: CGI-I Scale Score in LOCF Data.
Description: The efficacy of trial medication were rated for each participant using the Clinical Global Impression Improvement (CGI-I) scale. The study physician must rate the participant's total improvement whether or not it is due entirely to drug treatment. All responses were compared to the participant's condition a baseline. Response choices include: 0 = not assessed; 1 =very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 =minimally worse; 6 = much worse; and 7 = very much worse.
Time Frame: Week 1, 2 and 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Total: Participants were stabilized on one of the following atypical oral antipsychotic medication for at least 14 days before Day 1: risperidone, quetiapine, olanzapine, ziprasidone, or paliperidone. On Day 1, participants were administered a single aripiprazole IM depot 400 mg injection. Concomitant to the aripiprazole IM depot injection, participants continued to receive their current atypical antipsychotic medication for 14 days.
Arm/Group | Total
Number analyzed (Participants) | 60
Units on a scale
  Week 1 (N= 59) | 3.85 (0.45)
  Week 2 (N= 59) | 3.69 (0.56)
  Week 4 (N= 59) | 3.58 (0.77)

ADVERSE EVENTS:
Time Frame: From the time the ICF was signed until follow-up at 30 days after the last trial visit (Day 28).
Description: SAE was any untoward medical occurrence that resulted in death, life-threatening, required inpatient hospitalization or prolonged hospitalization. AE was an exacerbation of an existing problem, any new problem, experienced by a participant in a trial, whether or not considered drug related by study physician.
Arm/Group | Aripiprazole IM Depot 400mg
Serious Adverse Events (participants affected / at risk) | 1/60
Other Adverse Events (participants affected / at risk) | 35/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole IM Depot 400mg (N=60)
Suicide Attempt (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole IM Depot 400mg (N=60)
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Salivary hypersecretion (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 3
Injection site pain (General disorders) | 4
Irritability (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 1
Heart rate increased (Investigations) | 1
Weight increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Akathisia (Nervous system disorders) | 2
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dystonia (Nervous system disorders) | 3
Extrapyramidal disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Impatience (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Restlessness (Psychiatric disorders) | 3
Proteinuria (Renal and urinary disorders) | 1
Pyuria (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No